CLINICAL TRIAL: NCT06703437
Title: A Phase I Open Label Peri-prostatic Neuraxial Block With Lidocaine and Ethanol in High-risk Localized Prostate Cancer
Brief Title: Long Acting Neuraxial Peri-prostatic Block in Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Ali Zahalka, Clinical Instructor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-22-00221
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Long-acting neuraxial blockade (Experimental): Long-acting neuraxial blockade at the time of prostate biopsy by periprostatic injection of Dehydrated alcohol + lidocaine.
  Interventions: Drug: Dehydrated alcohol; Drug: Lidocaine IV

INTERVENTIONS:
Drug: Dehydrated alcohol — Long-acting neuraxial blockade at the time of prostate biopsy by periprostatic injection of Dehydrated alcohol.
Drug: Lidocaine IV — By periprostatic injection, 2mL

SUMMARY:
Disease progression after definitive therapy for prostate cancer is a major source of morbidity and mortality. Adrenergic/sympathetic innervation of the prostate is essential for prostate cancer progression, and abrogation of these signals by blocking adrenergic innervation halts disease progression. Long-acting neuraxial block of the sympathetic nerves that innervate the pelvis with dehydrated alcohol (>98% Ethanol) is a safe and effective tool in the treatment of chronic pelvic pain and cancer- induced pelvic pain. Furthermore, ultrasound guided periprostatic neuraxial block at the time of prostate biopsy with short-acting lidocaine is standard of care. Herein the research team proposes to administer a long-acting periprostatic neuraxial block with dehydrated alcohol and lidocaine under trans rectal ultrasound guidance in patients with high-risk clinical features for prostate cancer at the time of prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* PSA >10
* PSAD >0.15
* PI-RADS 5 lesion on MRI
* Karnofsky performance status >80
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Prior or concomitant treatment for prostate cancer, including radiation therapy, focal therapy, cryo therapy, androgen deprivation therapy.
* Imaging or clinical evidence of metastatic disease.
* PSA > 100ng/mL

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Limited to Male with high risk prostate cancer clinical features
Enrollment: 12 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | At week 2
  The DLT will be measured in the two week post administration period. The target toxicity rate is assumed as 25% considering immediate post-administration toxicity. This rate will not account for the delayed onset toxicities.
Maximally Tolerated Dose (MTD) | At week 2
  The MTD will be defined as the dose at which the isotonic estimate of the toxicity rate is closest to the target toxicity rate of 25%. The MTD will be used as a recommended dose for prospective Phase II study in future

SECONDARY OUTCOMES:
Time to biochemical recurrence | at month 6 and at year 2
  Absence or presence of any evidence of biochemical recurrence at two years after definitive treatment for prostate cancer.
Response Rate | at week 8
  Evidence of response supported by either histologic markers of treatment response, evidence based on difference in molecular proliferation markers between PBx and prostatectomy specimen.
Tumor immunogenicity | at week 8
  Evidence based on tumor immunogenicity as measured by PD1/PDL-1 expression by immunohistochemistry on final pathology.
Degree of neural inhibition | at week 8
  Histological quantification of adrenergic nerve density by tyrosine hydroxylase positive nerve staining

CONTACTS AND LOCATIONS:
Overall Officials: Ali Zahalka, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Ash Tewari, Study Director — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.
  To achieve aims in the approved proposal.
  Proposals should be directed to ali.zahalka@mountsinai.org. To gain access, data requestors need to sign a data access agreement. Proposals may be submitted up to 36 months following article publication. Data will be shared by email.